CLINICAL TRIAL: NCT05891782
Title: Effects of a HAPA-based Multicomponent Fall Intervention on Older Adults With Declines in Intrinsic Capacity in Nursing Homes
Brief Title: A HAPA-based Multicomponent Fall Intervention on Older Adults With Declines in Intrinsic Capacity in Nursing Homes
Acronym: HAPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZHANG Qing-hua (Other)
Responsible Party: Sponsor-Investigator, ZHANG Qing-hua, PhD, associate professor, Huzhou Normal University
Organization: Huzhou Normal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HuzhouU
Record Dates: First submitted 2023-05-16; First posted 2023-06-07 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Fall Risk
Keywords: Elderly; Nursing homes; Health behavior promotion

STUDY DESIGN:
Intervention Model Description: The study was planned as a randomized controlled clinical trial; by clustered randomization method, cases will be divided into two groups. There are 100 older adults in the nursing home to be studied. Study was planned as group 1 and group 2. The subjects will be assessed by blinded evaluators for primary and secondary outcomes at study baseline (T0), 4 weeks for the intention intervention (T1), 12 weeks for the action intervention (T2), and 8 weeks for the follow-up (T3).
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A HAPA-based multicomponent fall intervention will use group education, individualized plans and face-to-face interviews to develop health behaviors, such as fall emergency management, IC enhancement (exercise management, diet management, cognitive improvement, psychological regulation, vision protection), medication and disease management, environmental improvement, and fall self-efficacy enhancement.
  Interventions: Behavioral: HAPA-based Multidomain Fall Risk Management
- Control Group (Experimental): The control group will receive the same overall duration and frequency of interventions as the intervention group.
  Interventions: Behavioral: Regular health education lectures

INTERVENTIONS:
Behavioral: HAPA-based Multidomain Fall Risk Management — According to the HAPA and the conceptual model of IC, this intervention consists of 3 stages.
  Stage 1: The main format will be group lectures and scenario simulation, each intervention will have a duration of 30 to 45 minutes. Intervention content will utilize BCT [5.1, 5.3, 5.5, 5.6, 9.3, 15.1] .
  Stage 2: This stage will utilize mostly group lectures or one-to-one interviews, to provide an action and coping plan to participants for fall risk management. This will apply BCT [1.1-1.4, 4.1] at week 4.Firstly, individualized targets will be established. Secondly, professionals and participants will collaborate to develop an implementation plan.
  Stage 3:Recovery self-efficacy will be implemented as group discussions, with each intervention lasting 15-30 minutes. Maintenance will be implemented in one-to-one interviews, with each intervention lasting 15-30 minutes.Finally, the consolidation and outlook will provide the foundation for the habit formation of healthy behaviors.
  Other Names: HAPA-MFRM
  Arms: Intervention group
Behavioral: Regular health education lectures — Weeks 1-4 will be provided with fall-related regular health education lectures. Weeks 5-16 will have regular activities according to the daily arrangement of the nursing home. Meanwhile, telephone, WeChat, or face-to-face interviews will be conducted fortnightly, to understand the needs of the participants. During the process, staff will provide usual care such as vital signs monitoring, disease treatment, medication prescription, and health record maintenance.
  Other Names: Usual care
  Arms: Control Group

SUMMARY:
Falls are a common geriatric syndrome that impedes healthy aging and are the primary cause of accidental death in older adults. Globally, more than 50% of older adults experience falls in nursing homes each year. Intrinsic capacity (IC) is a quantifiable measure of healthy aging, and consists of five dimensions: cognitive, locomotor, vitality, sensory (vision and hearing), and psychological capacity. Decline in IC is an independent factor in the occurrence of falls in older adults. A related theoretical framework indicates that healthy behaviors are the key to enhance IC. The health action process approach (HAPA) has been shown to have positive effects on health behavior promotion. Therefore, the aim of this study is to examine the effect of multidimensional fall management based on HAPA on fall risk, fall efficacy, and healthy aging among older adults with declines in IC in Chinese nursing homes.

DETAILED DESCRIPTION:
Method： First, a randomly selected nursing home in Huzhou, will be selected for the study using the WHO Intrinsic Ability Screening Scale for older adults with declines in IC. A baseline assessment will be conducted followed by clustered randomization to divide into an intervention group (n=50) and a control group (n=50). All subjects will be intervened, after signing the informed consent. The subjects will be assessed by blinded evaluators for primary and secondary outcomes at at study baseline (T0), 4 weeks for the intention intervention (T1), 12 weeks for the action intervention (T2), and 8 weeks for the follow-up (T3). Finally, data collection and statistical processing will be carried out.

Expected results:

Reduce falls risk among the nursing home residents of the intervention group. Improvement of IG among the intervention group. Improvement of healthy aging among the intervention group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years.
2. Living in the nursing home for ≥ 3 months.
3. WHO screening tool identifies at least one dimension of decline in IC.
4. Ability to move independently (non-disabled) with a score of ≥ 4 on the SPPB.

(4) Voluntary involvement in the trial and informed consent provided by the participant.

Exclusion Criteria:

1. Have severe visual or hearing deprivation.
2. Have severe mental impairment or severe cognitive deficits (i.e., severe depression, schizophrenia).
3. Have severe and terminal heart, liver, brain, and kidney disease (i.e., tumors, brain trauma).
4. Other trials received within 6 months prior to the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Intrinsic capacity (IC) composite score | baseline, after 4 weeks, after 16 weeks, after 24 weeks
  Each dimension of capability will be assigned score of 1, so the composite score ranges from 0-5, with higher scores representing a decline in IC
The Mini-mental State Examination (MMSE) | baseline, after 4 weeks, after 16 weeks, after 24 weeks
  MMSE is a widely used assessment instrument with a score range of 0-30, and the Cronbach's alpha coefficient was 0.833 for internal consistency. Subject to age and culture, the normal thresholds are classified according to the education level, the classification criteria are: illiterate > 17, primary > 20, high school and above > 24 as cognitive normal.
The Short Physical Performance Battery (SPPB) | baseline, after 4 weeks, after 16 weeks, after 24 weeks
  SPPB as a recommended physical performance test, combines the balance test, the gait speed test, and the chair rise test. The total scores range from 0 (worst performance) to 12 (best performance), and the Cronbach's alpha coefficient was 0.76 for internal consistency.
The Mini-Nutritional Assessment (MNA) | baseline, after 4 weeks, after 16 weeks, after 24 weeks
  MNA is suitable for assessing the vitality of older people, covering anthropometric indicators, dietary and subjective assessments. The total score of the scale is 30, 24-30 is considered good nutritional status, 17-23.5 is at risk of malnutrition, and <17 is considered malnutrition. And the Cronbach's alpha coefficient was 0.71 for internal consistency.
Sensory capacity assessment | baseline, after 4 weeks, after 16 weeks, after 24 weeks
  Visual capacity will use the self-report (one item of the WHO ICOPE screening tool) format. If the participant denies visual impairment, a tumbling E chart will be used to standardize visual testing. According to the Standard for Logarithmic Visual Acuity Charts (GB11533-2011), the decimal record will be used. Hearing capacity will use the self-report (two items of the WHO ICOPE screening tool). If the participant denies hearing impairment, a whisper voice test will be used. The examiner will stand behind the participant at an arm's length (0.6 meters). The examiner will whisper common and unrelated four words, and the participant will be required to repeat the words.
The Patient Health Questionnaire-9 (PHQ-9) | baseline, after 4 weeks, after 16 weeks, after 24 weeks
  PHQ-9 will assess the frequency of nine depressive symptoms over the past two weeks. The scale has a total score range of 0-27, with scores of 5 and above considering observation or counseling. And the Cronbach's alpha coefficient was 0.82 for internal consistency.
The Self-Rated Fall Risk Questionnaire (SFRQ) | baseline, after 4 weeks, after 16 weeks, after 24 weeks
  FRQ was developed by the CDC, which contains 12 items totaling 14 scores, with a score of ≥4 suggesting a risk of falling, and the Cronbach's alpha coefficient was 0.724 for internal consistency.

SECONDARY OUTCOMES:
Timed-Up-and-Go Test (TUG) | baseline, after 16 weeks, after 24 weeks
  TUG assesses gait and balance in older adults. The participant will sit on the chair, and when the command "start" is heard, they will walk forward as fast as possible to 3 meters, then turn around and walk back to the chair.
Hand Grip Strength (HGS) | baseline, after 16 weeks, after 24 weeks
  HGS will be tested using a hand dynamometer (CAMRY). Participants will be required to rest for at least 1 minute before having their grip strength measured. Measurements will be taken in a seated position and dominant hand, with the elbow angle at 90° and the forearm in a neutral position. A maximal squeeze will be performed during the measurement, maintaining body posture, and averaged over three times.
The Modified Falls Efficacy Scale (MFES) | baseline, after 4 weeks, after 16 weeks, after 24 weeks
  MFES was revised in 1996 by Keith Hill et al . The scale is suitable for measuring FOF and activity balance confidence. It consists of 14 items (9 indoor activities and 5 outdoor activities), each of which can be selected on a scale of 0-10, and the Cronbach's alpha coefficient was 0.974 for internal consistency.
The self-management abilities for fall prevention in elderly questionnaire | baseline, after 4 weeks, after 16 weeks, after 24 weeks
  It was developed by Huang et al in 2017. The questionnaire contains 7 dimensions with 42 items, the total score ranges from 42 to 210, and the Cronbach's alpha coefficient of the questionnaire is 0.775.
The Fall Management Behavior Change Stage Assessment | baseline, after 4 weeks, after 16 weeks, after 24 weeks
  It was developed based on Lippke et al. This scale consists of only one entry: Do you follow the principles of "appropriate exercise, proper diet, emotional adjustment, cognitive improvement, visual and auditory improvement, management of illness and medication, and environmental screening" for fall risk management? Participants selected "No, I have no intention to start falls risk management at this time" for the pre-intention stage; "No, but I have decided to start falls risk management" for the intention stage; and "Yes" for the action stage. The scale had a retest reliability of 0.851.
The Healthy Aging Instrument (HAI) | baseline, after 16 weeks, after 24 weeks
  The scale covers 9 domains: living a sufficient and simple life, acceptance of aging, stress management, having social relationships and support, helping others, self-care, normal physical functioning, normal cognitive functioning, and social participation. The 35-item scale has a total score of 35-175, with higher scores indicating better levels of healthy aging.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghua Zhang, PhD, Principal Investigator — School of Medicine & Nursing Sciences, Huzhou University
Locations (1):
- Huzhou Social Welfare Center, Huzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beard JR, Officer AM, Cassels AK. The World Report on Ageing and Health. Gerontologist. 2016 Apr;56 Suppl 2:S163-6. doi: 10.1093/geront/gnw037. No abstract available. PMID 26994257
- [Background] Zhou Y, Ma L. Intrinsic Capacity in Older Adults: Recent Advances. Aging Dis. 2022 Apr 1;13(2):353-359. doi: 10.14336/AD.2021.0818. eCollection 2022 Apr. PMID 35371613
- [Background] Chhetri JK, Xue QL, Ma L, Chan P, Varadhan R. Intrinsic Capacity as a Determinant of Physical Resilience in Older Adults. J Nutr Health Aging. 2021;25(8):1006-1011. doi: 10.1007/s12603-021-1629-z. PMID 34545921
- [Background] Schwarzer R, Lippke S, Luszczynska A. Mechanisms of health behavior change in persons with chronic illness or disability: the Health Action Process Approach (HAPA). Rehabil Psychol. 2011 Aug;56(3):161-70. doi: 10.1037/a0024509. PMID 21767036
- [Background] Treacy D, Hassett L. The Short Physical Performance Battery. J Physiother. 2018 Jan;64(1):61. doi: 10.1016/j.jphys.2017.04.002. Epub 2017 Jun 20. No abstract available. PMID 28645532
- [Background] Vellas B, Guigoz Y, Garry PJ, Nourhashemi F, Bennahum D, Lauque S, Albarede JL. The Mini Nutritional Assessment (MNA) and its use in grading the nutritional state of elderly patients. Nutrition. 1999 Feb;15(2):116-22. doi: 10.1016/s0899-9007(98)00171-3. PMID 9990575
- [Background] Xia NG, Lin JH, Ding SQ, Dong FR, Shen JZ, Du YR, Wang XS, Chen YY, Zhu ZG, Zheng RY, Xu HQ. Reliability and validity of the Chinese version of the Patient Health Questionnaire 9 (C-PHQ-9) in patients with epilepsy. Epilepsy Behav. 2019 Jun;95:65-69. doi: 10.1016/j.yebeh.2019.03.049. Epub 2019 Apr 24. PMID 31026785
- [Background] Lach HW, Ball LJ, Birge SJ. The Nursing Home Falls Self-Efficacy Scale: development and testing. Clin Nurs Res. 2012 Feb;21(1):79-91. doi: 10.1177/1054773811426927. Epub 2011 Oct 31. PMID 22042908
- [Background] Thanakwang K, Soonthorndhada K. Mechanisms by which social support networks influence healthy aging among Thai community-dwelling elderly. J Aging Health. 2011 Dec;23(8):1352-78. doi: 10.1177/0898264311418503. Epub 2011 Aug 23. PMID 21862701
- [Background] Tinetti ME. Performance-oriented assessment of mobility problems in elderly patients. J Am Geriatr Soc. 1986 Feb;34(2):119-26. doi: 10.1111/j.1532-5415.1986.tb05480.x. No abstract available. PMID 3944402
- [Derived] Shang S, Cheng S, Qi L, Liu T, Yang Y, Yao X, Lu D, Cheng X, Yang J, Cheng M, Zhang Q. Effectiveness of HAPA-based multidomain fall risk management for older adults with declining intrinsic capacity in nursing homes: protocol of a randomised controlled trial. BMJ Open. 2025 Apr 30;15(4):e082702. doi: 10.1136/bmjopen-2023-082702. PMID 40306996